CLINICAL TRIAL: NCT01136850
Title: Intermittent Preventive Treatment With Azithromycin-containing Regimens for the Prevention of Malarial Infections and Anaemia and the Control of Sexually Transmitted Infections in Pregnant Women in Papua New Guinea
Brief Title: Intermittent Preventive Treatment With Azithromycin-containing Regimens in Pregnant Women in Papua New Guinea
Acronym: IPTp in PNG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: Papua New Guinea Institute of Medical Research (Other Government); The University of Western Australia (Other); Walter and Eliza Hall Institute of Medical Research (Other); University of Barcelona (Other)
Responsible Party: Principal Investigator, Stephen Rogerson, Professor of Medicine, University of Melbourne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 70270
Record Dates: First submitted 2010-04-06; First posted 2010-06-04 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Malaria in Pregnancy; Sexually Transmitted Infections; Anaemia
Keywords: Plasmodium falciparum; Plasmodium vivax; azithromycin; sulphadoxine pyrimethamine; low birth weight; haemoglobin; Chlamydia trachomatis; Neisseria gonorrhoeae; Treponema pallidum
MeSH Terms: conditions — Sexually Transmitted Diseases; Anemia; Malaria, Falciparum; Malaria, Vivax; Treponemal Infections | interventions — Chloroquine; fanasil, pyrimethamine drug combination; Azithromycin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SP, chloroquine treatment; bed net (Active Comparator): Treatment course of sulphadoxine pyrimethamine and chloroquine on enrolment. Long lasting insecticide treated bed net
  Interventions: Drug: chloroquine, sulphadoxine pyrimethamine, LLIN
- 3 x SP plus azithromycin; bed nets (Experimental): Three x monthly courses of azithromycin and sulphadoxine pyrimethamine plus long lasting insecticide treated bed net.
  Interventions: Drug: azithromycin, sulphadoxine pyrimethamine, LLIN

INTERVENTIONS:
Drug: chloroquine, sulphadoxine pyrimethamine, LLIN — > 50Kg: chloroquine base 150 mg 4 tablets daily for 3 days, plus sulphadoxine pyrimethamine 1500/75 mg single dose.
  < 50 Kg: chloroquine base 150 mg 3 tablets daily for 3 days, plus sulphadoxine pyrimethamine 1500/75 mg single dose.
  Given at enrolment, 14-26 weeks gestation, by mouth.
  Other Names: sulfadoxine-pyrimethamine
  Arms: SP, chloroquine treatment; bed net
Drug: azithromycin, sulphadoxine pyrimethamine, LLIN — sulphadoxine pyrimethamine (1500 mg/75 mg as single dose) plus azithromycin (1 g twice daily for 2 days).
  Given three times by mouth at monthly intervals, commencing at between 14 and 26 weeks gestation.
  Other Names: Zithromax; sulfadoxine-pyrimethamine
  Arms: 3 x SP plus azithromycin; bed nets

SUMMARY:
The purpose of this study is to determine whether repeated courses of sulphadoxine-pyrimethamine (SP) in combination with azithromycin given at Antenatal Clinic, leads to lower rates of low birth weight deliveries (<2.5 kg) among Papua New Guinean women, than the current standard treatment of SP and chloroquine.

ELIGIBILITY:
Inclusion Criteria:

* pregnant
* 14-26 weeks'gestation
* permanent resident of study area
* exclusive use of study health facilities for primary health care
* Age is between 16 and 49 years

Exclusion Criteria:

* Known chronic illness, e.g. TB, diabetes, renal failure
* Severe anaemia requiring hospitalisation (Hb < 6 g/dl accompanied by symptoms requiring urgent treatment)
* permanent disability, that prevents or impedes study participation and/or comprehension
* Known multiple pregnancy

Ages: 16 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2793 (Actual)
Dates: Start 2009-11; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Proportion of women delivering low birth weight babies, <2500 g | At delivery

SECONDARY OUTCOMES:
Prevalence of P falciparum at delivery in peripheral, placental and cord blood films and on placental histology | at delivery
Mean maternal hemoglobin concentration at delivery, and proportion of women anaemic (Hb < 11 g/dl). | At delivery
Prevalence (at enrolment, second treatment, and delivery) and consequences (maternal haemoglobin, birth weight and placental pathology) of P. vivax infection in pregnancy | up to 26 weeks
  From enrolment at 14-26 weeks gestation, until delivery
Incidence of symptomatic malaria during pregnancy | Up to 26 weeks
  From enrolment at 14-26 weeks until delivery
Proportion of women carrying azithromycin-sensitive sexually transmitted infections at second treatment visit (28-34 weeks). | 28-34 week gestation study visit
Incidence of Adverse Events, including severe adverse events (SAEs), and AEs possibly or probably associated with study medications | 14-26 weeks
  From enrolment at 14-26 weeks gestation until delivery
Prevalence of drug resistance markers in parasites infecting women in late pregnancy, particularly in the P falciparum and P vivax dihydrofolate reductase and dihydropteroate synthase enzymes, associated with SP resistance | at delivery
Prevalence and antibiotic sensitivity patterns of S. pneumoniae in nasopharyngeal swabs collected at delivery | at delivery
Maternal, perinatal and infant mortality rates | Mothers; up to 32 weeks, from enrolment at 14-26 weeks gestation, until delivery. Pernatal: 16 weeks, from 28 weeks gestation to 4 weeks of age. Infant: from live birth to 1 year of age
  maternal mortality is during pregnancy and until 6 weeks post partum. Perinatal mortality is from 28 weeks gestation until 6 weeks postpartum. Infant mortality is from irth to 12 months of age
Impact of IPTp on development of immunity to malaria in pregnancy | at delivery
Characteristics of parasites infecting pregnant women | Up to 26 weeks, from 14-26 weeks gestation until delivery

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Rogerson, FRACP PhD, Principal Investigator — University of Melbourne
Locations (1):
- Papua New Guinea Institute of Medical Research, Madang, Madang Province, Papua New Guinea

REFERENCES:
- [Background] Steketee RW, Nahlen BL, Parise ME, Menendez C. The burden of malaria in pregnancy in malaria-endemic areas. Am J Trop Med Hyg. 2001 Jan-Feb;64(1-2 Suppl):28-35. doi: 10.4269/ajtmh.2001.64.28. PMID 11425175
- [Background] Guyatt HL, Snow RW. The epidemiology and burden of Plasmodium falciparum-related anemia among pregnant women in sub-Saharan Africa. Am J Trop Med Hyg. 2001 Jan-Feb;64(1-2 Suppl):36-44. doi: 10.4269/ajtmh.2001.64.36. PMID 11425176
- [Background] Brabin B, Piper C. Anaemia- and malaria-attributable low birthweight in two populations in Papua New Guinea. Ann Hum Biol. 1997 Nov-Dec;24(6):547-55. doi: 10.1080/03014469700005312. PMID 9395740
- [Background] Benet A, Khong TY, Ura A, Samen R, Lorry K, Mellombo M, Tavul L, Baea K, Rogerson SJ, Cortes A. Placental malaria in women with South-East Asian ovalocytosis. Am J Trop Med Hyg. 2006 Oct;75(4):597-604. PMID 17038679
- [Background] Allen SJ, Raiko A, O'Donnell A, Alexander ND, Clegg JB. Causes of preterm delivery and intrauterine growth retardation in a malaria endemic region of Papua New Guinea. Arch Dis Child Fetal Neonatal Ed. 1998 Sep;79(2):F135-40. doi: 10.1136/fn.79.2.f135. PMID 9828741
- [Background] Schultz LJ, Steketee RW, Macheso A, Kazembe P, Chitsulo L, Wirima JJ. The efficacy of antimalarial regimens containing sulfadoxine-pyrimethamine and/or chloroquine in preventing peripheral and placental Plasmodium falciparum infection among pregnant women in Malawi. Am J Trop Med Hyg. 1994 Nov;51(5):515-22. doi: 10.4269/ajtmh.1994.51.515. PMID 7985742
- [Background] Parise ME, Ayisi JG, Nahlen BL, Schultz LJ, Roberts JM, Misore A, Muga R, Oloo AJ, Steketee RW. Efficacy of sulfadoxine-pyrimethamine for prevention of placental malaria in an area of Kenya with a high prevalence of malaria and human immunodeficiency virus infection. Am J Trop Med Hyg. 1998 Nov;59(5):813-22. doi: 10.4269/ajtmh.1998.59.813. PMID 9840604
- [Background] Verhoeff FH, Brabin BJ, Chimsuku L, Kazembe P, Russell WB, Broadhead RL. An evaluation of the effects of intermittent sulfadoxine-pyrimethamine treatment in pregnancy on parasite clearance and risk of low birthweight in rural Malawi. Ann Trop Med Parasitol. 1998 Mar;92(2):141-50. doi: 10.1080/00034989859979. PMID 9625909
- [Background] Shulman CE, Dorman EK, Cutts F, Kawuondo K, Bulmer JN, Peshu N, Marsh K. Intermittent sulphadoxine-pyrimethamine to prevent severe anaemia secondary to malaria in pregnancy: a randomised placebo-controlled trial. Lancet. 1999 Feb 20;353(9153):632-6. doi: 10.1016/s0140-6736(98)07318-8. PMID 10030329
- [Background] Casey GJ, Ginny M, Uranoli M, Mueller I, Reeder JC, Genton B, Cowman AF. Molecular analysis of Plasmodium falciparum from drug treatment failure patients in Papua New Guinea. Am J Trop Med Hyg. 2004 Mar;70(3):251-5. PMID 15031512
- [Background] ter Kuile FO, van Eijk AM, Filler SJ. Effect of sulfadoxine-pyrimethamine resistance on the efficacy of intermittent preventive therapy for malaria control during pregnancy: a systematic review. JAMA. 2007 Jun 20;297(23):2603-16. doi: 10.1001/jama.297.23.2603. PMID 17579229
- [Background] Kalilani L, Mofolo I, Chaponda M, Rogerson SJ, Alker AP, Kwiek JJ, Meshnick SR. A randomized controlled pilot trial of azithromycin or artesunate added to sulfadoxine-pyrimethamine as treatment for malaria in pregnant women. PLoS One. 2007 Nov 14;2(11):e1166. doi: 10.1371/journal.pone.0001166. PMID 18000538
- [Derived] Unger HW, Bleicher A, Ome-Kaius M, Aitken EH, Rogerson SJ. Associations of maternal iron deficiency with malaria infection in a cohort of pregnant Papua New Guinean women. Malar J. 2022 May 26;21(1):153. doi: 10.1186/s12936-022-04177-8. PMID 35619134
- [Derived] Unger HW, Laurita Longo V, Bleicher A, Ome-Kaius M, Karl S, Simpson JA, Karahalios A, Aitken EH, Rogerson SJ. The relationship between markers of antenatal iron stores and birth outcomes differs by malaria prevention regimen-a prospective cohort study. BMC Med. 2021 Oct 5;19(1):236. doi: 10.1186/s12916-021-02114-1. PMID 34607575
- [Derived] Aitken EH, Damelang T, Ortega-Pajares A, Alemu A, Hasang W, Dini S, Unger HW, Ome-Kaius M, Nielsen MA, Salanti A, Smith J, Kent S, Hogarth PM, Wines BD, Simpson JA, Chung AW, Rogerson SJ. Developing a multivariate prediction model of antibody features associated with protection of malaria-infected pregnant women from placental malaria. Elife. 2021 Jun 29;10:e65776. doi: 10.7554/eLife.65776. PMID 34181872
- [Derived] Ome-Kaius M, Karl S, Wangnapi RA, Bolnga JW, Mola G, Walker J, Mueller I, Unger HW, Rogerson SJ. Effects of Plasmodium falciparum infection on umbilical artery resistance and intrafetal blood flow distribution: a Doppler ultrasound study from Papua New Guinea. Malar J. 2017 Jan 19;16(1):35. doi: 10.1186/s12936-017-1689-z. PMID 28103875
- [Derived] Ome-Kaius M, Unger HW, Singirok D, Wangnapi RA, Hanieh S, Umbers AJ, Elizah J, Siba P, Mueller I, Rogerson SJ. Determining effects of areca (betel) nut chewing in a prospective cohort of pregnant women in Madang Province, Papua New Guinea. BMC Pregnancy Childbirth. 2015 Aug 19;15:177. doi: 10.1186/s12884-015-0615-z. PMID 26286026
- [Derived] Teo A, Hasang W, Randall LM, Unger HW, Siba PM, Mueller I, Brown GV, Rogerson SJ. Malaria preventive therapy in pregnancy and its potential impact on immunity to malaria in an area of declining transmission. Malar J. 2015 May 26;14:215. doi: 10.1186/s12936-015-0736-x. PMID 26006260
- [Derived] Unger HW, Ome-Kaius M, Wangnapi RA, Umbers AJ, Hanieh S, Suen CS, Robinson LJ, Rosanas-Urgell A, Wapling J, Lufele E, Kongs C, Samol P, Sui D, Singirok D, Bardaji A, Schofield L, Menendez C, Betuela I, Siba P, Mueller I, Rogerson SJ. Sulphadoxine-pyrimethamine plus azithromycin for the prevention of low birthweight in Papua New Guinea: a randomised controlled trial. BMC Med. 2015 Jan 16;13:9. doi: 10.1186/s12916-014-0258-3. PMID 25591391
- See also: home page of umbrella organisation coordinating this and other trials on malaria in pregnancy — http://mip-consortium.org
- See also: home page of Department of Central contact person, Dr Rogerson — http://www.medrmhwh.unimelb.edu.au/
- See also: home page of Papua New Guinea Institute of Medical Research — http://www.pngimr.org.pg